CLINICAL TRIAL: NCT04834648
Title: Operations Research to Improve Timely Referral Flow and Compliance of Diabetic Retinopathy Patients From Peripheral Eye Care Centers to Tertiary Center in Nepal: Cluster Randomised Control Trial
Brief Title: Improve Timely Referral Flow and Compliance of Diabetic Retinopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seva Foundation (Other)
Collaborators: Lumbini Eye Institute and Research Centre (Other); Indian Institute of Public Health, India (Other); Seva Canada Society (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LEI/IRC/09/019/20
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Diabetes; Diabetic Retinopathy
Keywords: referral rate; diabetic retinopathy; counselling
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: At LEI the staff will be blinded about the intervention/ control referring centers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Counseling (Experimental): Structured Counseling, which includes A. Counseling is done by a trained counselor
  B. Telephonic Follow up:
  C. Development of Fast Track system at the Base Hospital. D. Provide Health Education Material to all Diabetic Patients. E. Referral communication and feedback between referring and referral facility.
  Interventions: Behavioral: Structured Counseling
- Control Arm (No Intervention): General Counseling, which included saying you need to visit the hospital and you have involvement in the eyes due to diabetes, providing a health education leaflet.

INTERVENTIONS:
Behavioral: Structured Counseling — Structured Counseling, which includes A. Counseling is done by a trained counselor
  B. Telephonic Follow up:
  C. Development of Fast Track system at the Base Hospital. D. Provide Health Education Material to all Diabetic Patients. E. Referral communication and feedback between referring and referral facility.
  Arms: Structured Counseling

SUMMARY:
An effective referral system helps to ensure a close relationship between all levels of the health system and ensures clients receive optimum care at the appropriate level and at affordable cost, and hospital facilities are used optimally and cost-effectively. A referral system requires consideration of all its important components that can be then adjusted to the local situation. Being a system, the important components of a referral system are Health system issues (Service providers, Referral protocols, Communication & transportation provide), Referring facility& Referral practicalities (Client & their condition, Protocols of care, Care provider & documents, Referral decision, Outward referral form, Communicate with referral facility, Client information, Referral register), Referral facility& Referral practicalities (Client with referral form, Treat the client with the document, Rehabilitation plan, Back referral form, Feedback to referring facility, Referral register) and Supervision and capacity building (Referral monitoring, Ensure back referral, Feedback and training to facility staff and Feedback to central level) ((USAID), 2012).

There are mainly two limitations on referring Diabetic Retinopathy patients. Patient-related reasons: lack of awareness, belief, cost, distance from screening/ treatment centers, discomfort from dilating drops, efforts to attend yet another center, fear of laser treatment, fear of its impact on quality of life and jobs, lack of family support and guilt surrounding the failure to control blood sugar. Provider-related reasons are poor counseling and advisory services about ocular complications for patients with diabetes, inefficient call and recall system, long waiting times for screening or treatment, and complicated referral mechanism.

Lumbini eye institute is a comprehensive tertiary eye care center in western Nepal. In spite of 19 peripheral referral centers under it, there is a poor inflow of Diabetic retinopathy patients as against the estimated disease burden in the catchment area. The objective of our study is to improve timely referral flow from referring centers and compliance with referral cases after the intervention. In order to meet our objective, the investigators tend to implement patient counseling at referral centers, a referral tracking system, and a fast-track mechanism for patients at base hospitals.

DETAILED DESCRIPTION:
Background: Changes in lifestyle and a growing number of aging populations have increased the prevalence of diabetes worldwide. Diabetes imposes a heavy disease burden in both developed and developing countries (1). Diabetic retinopathy is the commonest microvascular complication of diabetes and the leading cause of blindness in adults. There are no symptoms initially; visual impairment is seen in the proliferative stage and in macular involvement. Vision once lost will never be regained (2). The prevalence of diabetic retinopathy was 10%-50% for Type 1 and 25.2% for Type2. The worldwide prevalence of diabetic retinopathy was found to be 34.6%. WHO estimates Diabetic retinopathy is responsible for 4.8% of 37 million cases of blindness throughout the world. Several studies in Nepal showed the prevalence of 9% to 78%. A study at LEIRC showed PDR and ADED to 34%; this suggests a major blockage of cases at the tertiary and primary level (2013-2014).

Early diagnosis and treatment are the key components to reduce Diabetic blindness. A comprehensive set of guidelines (CARE 2019) recommends initial dilatation and comprehensive eye examination by an optometrist or ophthalmologist. Patient with Mild, Moderate and Severe Diabetic retinopathy requires a referral and they need reexamination or follow up within time limit of 3-6 months, less than 3 months and less than 1 month respectively. Incidence of visual loss secondary to proliferative Diabetic Retinopathy can be reduced by referral to an ophthalmologist. Multiple studies show laser photocoagulation of new vessels reduces the incidence of Diabetic Blindness by 60% to 80%.

Lumbini eye institute is a comprehensive tertiary eye care center in western Nepal. In spite of 19 peripheral referral centers under it, there is a poor inflow of Diabetic retinopathy patients as against the estimated disease burden in the catchment area. There are mainly two limitations on referring Diabetic Retinopathy patients. Patient-related reasons: lack of awareness, belief, cost, distance from screening/ treatment centers, discomfort from dilating drops, efforts to attend yet another center, fear of laser treatment, fear of its impact on quality of life and jobs, lack of family support and guilt surrounding the failure to control blood sugar. Provider-related reasons are poor counseling and advisory services about ocular complications for patients of diabetes, inefficient call and recall system, long waiting times for screening or treatment, and complicated referral mechanism (2). Considering these reasons and problem tree analysis effective interventions designed. Counseling and telephonic follow-up at referring facility; fast track system at the base hospital. The objective of our study is to improve timely referral flow from referring centers and compliance with referral cases after the intervention.

Methods:

Study Design: Two arm parallel, cluster Randomised control trial with allocation ratio 1:1 will be used.

Study Setting :

All diabetic retinopathy patients attending peripheral eye care centers will be the study population.

Lumbini Eye Institute and Research Center (LEIRC) - a comprehensive tertiary referral eye care center located in the Western part of Nepal has nineteen referring centers: five secondary eye hospitals (SEC), three district eye care centers (DECC), and eleven primary eye care centers (PECC). The referral center (LEIRC) has several sub-specialty services; the Retina department is well equipped with two consultants, one retina fellow, and one separate counselor. A secondary eye hospital has a general ophthalmologist, ophthalmic paramedical personnel (optometrist/ophthalmic assistant), and a counselor with limited diagnostic tools for diabetic retinopathy (DR). A primary/district eye care center has ophthalmic paramedical personnel (optometrist/ophthalmic assistant) and an optician with a direct ophthalmoscope for retina examination.

Masking: At LEI the staff will be blinded about the intervention/ control referring centers.

Data collection plan: An experienced team member will be responsible for data collection and telephonic follow-up. the project coordinator will be trained thoroughly trained on the completion of the data collection form Data Management Plan: The demographic information and other variables of the patient who are referred from peripheral eye care centers will be collected and entered in an excel sheet. One of the team members will be responsible for data management.

Data Analytic plan: Data will be analyzed using IBM SPSS. Differences indifference in compliance and referral rates will be computed.

Study period: Approximately 19 months (March 2020 to December 2021) Ethical consideration: Ethical approval is taken from the Institutional review committee, LEIRC. Data confidentiality will be maintained.

Ethical considerations:

Written Consent form including the title of the study and their support during the study period was sent to all 10 centers included in the study. These consent forms were signed by the head of centers on 12th June 2020 and sent to LEIRC. Ethical Approval from the Institutional Review Committee (IRC) of LEIRC was taken on 8th August 2020. Data confidentiality will be maintained. No personal information will be used in analysis, reports, and publications.

Discussion:

Diabetic Retinopathy is a global epidemic in both developed and developing countries with significant morbidity and mortality. In a study done by Mishra SK et al, they found people were less aware of the microvascular complications of diabetes. They didn't meet the physician regularly for diabetes control and didn't know about regular eye examinations with ophthalmologists. Even though the incidence of blindness secondary to diabetes mellitus can be significantly reduced; there is still a large number of diabetes patient with vision loss due to retinal complications of the disease In a study done by Tien Y. Wang et al, they came with a broad-based system-level approach to prevent vision loss resulting from Diabetic Retinopathy: 1: Targeted health care education to improve public knowledge. 2: well-implemented community or national level screening programs for all patients with diabetes. 3: Timely referral for severe level of Diabetic Retinopathy. 4: Appropriate treatment for advanced Diabetic Retinopathy (PDR and DME).

In our study the investigators wanted to make the patient aware of the changes diabetes can bring to the eye, the investigators implemented Structured Counseling where the patient is explained in detail about the changes diabetes makes in the eye. It also includes the impact on vision and different treatment options available and the rate. They are also explained to go to a base hospital where they will be evaluated by a retina specialist thus decreasing a load of visual impairment due to diabetes.

World Health Organization (WHO) has identified adherence to follow-up services as a key component in effective management of Diabetic Retinopathy9. In this study, they found improving the clarity of the referral process by explaining the treatment costs, the reason for referral, and likely health benefits to the patient helped by increasing follow-up rates9. Keeping this in the investigators explained the treatment cost and about the base hospital in detain as our structured counseling. A study done by Mishra SK et al found major facilitator was the existence of referral slips to expedite treatment upon reaching the health facility and the major barrier was a failure to receive preferential treatment at the facility, despite the presence of the slip. In addition to this, they found lack of feedback as a barrier to functional referral system 3.

Similarly, during our problem tree analysis, the investigators found a longer waiting time and no preferential treatment as a factor in the referral system. The investigators tried implementing a referral slip and planned to decrease the waiting time by allowing them to visit the ophthalmologist directly at our center. This point will also be explained by the counselor during counseling.

ELIGIBILITY:
Inclusion Criteria:

* All Diabetic Retinopathy patients attending the peripheral eye centers linked with LEIRC.

Exclusion Criteria:

* All referred Diabetic patients who not is willing to be part of the study.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 8 months
  Percentage of referral compliance before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Lumbini Eye Institute and Research Center, Butwāl, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhattarai B, Thapa HB, Bashyal S, Thapa SK, Chaudhuri S, Agiwal V, Pant H, Singh S, Mahajan H. Structured Counselling and Regular Telephonic follow up to improve Referral flow and compliance in Nepal for Diabetic Retinopathy(SCREEN-D Study): a randomised controlled trial. BMC Health Serv Res. 2024 Feb 10;24(1):188. doi: 10.1186/s12913-024-10647-3. PMID 38336691